CLINICAL TRIAL: NCT00297310
Title: Pre-transplant Pharmacokinetics as a Predictor of the Tacrolimus Dose Requirement Post Renal Transplantation
Brief Title: Pre-transplant Assessment of Tacrolimus Blood Level Concentration, as a Predictor of Tacrolimus Dose Requirements After Kidney Transplantation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen-Cilag Pty Ltd (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR005020
Record Dates: First submitted 2006-02-24; First posted 2006-02-28 (Estimated); Last update posted 2011-06-20 (Estimated); Status verified 2010-04

CONDITIONS: Kidney Transplantation; Transplantation
Keywords: Tacrolimus; Kidney transplantation; Transplantation; Kidney failure; chronic; P-Glycoprotein
MeSH Terms: conditions — Renal Insufficiency; Bronchiolitis Obliterans Syndrome | interventions — Tacrolimus

INTERVENTIONS:
Drug: tacrolimus

SUMMARY:
The purpose of this study is to evaluate two groups of kidney transplant recipients, to determine the proportion of patients that achieve therapeutic blood concentrations of tacrolimus by Day 3 after transplantation. Patients in one group will be treated with tacrolimus according current clinical practice. The other group will have a pre-transplant assessment of their tacrolimus blood level concentration that will be used to guide post-transplantation tacrolimus dosing. Tacrolimus is a medicine that slows down the body's immune system. For this reason, it works as an anti-rejection medicine.

DETAILED DESCRIPTION:
This study is a multicentre, open-label, prospective, 2-arm, phase IV study of tacrolimus in renal transplant recipients. Patients will be randomized to receive current clinical practice or to have a pre-transplant pharmacokinetic assessment of tacrolimus metabolism that will be used to guide post-transplantation tacrolimus dosing, with the aim of increasing the proportion of patients that achieve a tacrolimus whole blood trough level of >10 ng/mL by Day 3 post-transplantation. Patients randomized to Group 1 will take a single dose of tacrolimus (0.1 mg/kg) prior to transplantation and a blood sample will be taken to determine tacrolimus whole blood concentration at 2 hours post-dose. The result of this blood sample will be used to guide tacrolimus dosing post-transplantation. Patients that return a low tacrolimus blood concentration will have a post-transplantation starting dose of up to 0.3 mg/kg/day, whereas patients that return a high tacrolimus blood concentration will have a post-transplantation starting dose of 0.1 mg/kg/day. Patients randomized to Group 2 will also receive a single pre-operative dose of tacrolimus, but will not have their tacrolimus whole blood concentration measured at 2 hours post-dose. These patients will be managed as per standard care.

The primary objective of the trial is to compare, between the two groups, the proportion of patients that achieve a tacrolimus whole blood trough concentration of ³10 ng/mL by Day 3 post-transplantation. The hypothesis is that performing a tacrolimus whole blood concentration assessment 2 hours after a pre-operative dose (to guide tacrolimus dosing post-transplantation), will lead to an increase in the numbers of patients that achieve therapeutic blood concentrations post-transplant. The tacrolimus whole blood concentration at Day 3 post-transplantation is a marker of the risk of rejection and toxicity.

A substudy is being conducted which seeks to examine and compare clinical variability in absorption profile by measurement of the phenotype (blood levels) in kidney transplant recipients and determine the nature and extent of relationship with MDR-1 genotype, thus allowing the most predictive and cost effective method of determining tacrolimus dosing.

Pre-transplant: One single tacrolimus dose 0.1 mg/kg/day orally. Post-transplant: 0.15 - 0.3 mg/kg/day as two divided tacrolimus doses orally, the actual dose to be guided by the pre-transplant tacrolimus blood concentration.

ELIGIBILITY:
Inclusion Criteria:

* Patient has end-stage kidney disease and is a suitable candidate for primary renal transplantation or re-transplantation
* Patient is receiving a kidney transplant from a cadaveric or living (not HLA identical) donor, at least 10 years of age, with compatible ABO blood type

Exclusion Criteria:

* Patients receiving a graft from a non-heart-beating donor
* known to have significant liver disease, or is receiving a graft from a hepatitis C or B positive donor
* previously received or is receiving an organ transplant other than a kidney
* taking diltiazem, or any of the other disallowed medications during the 7 days prior to, and the 30 day trial period, or has been taking an investigational drug in the past 28 days
* patient or donor known to be HIV positive

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2004-05; Primary Completion 2006-10 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
The proportion of patients that achieve a tacrolimus whole blood trough concentration of >=10 ng/mL by Day 3 post-transplantation

SECONDARY OUTCOMES:
Time to achieve first trough concentration of >=10 ng/mL. Comparative number of dose changes in each arm post-transplantation. Number of patients with whole blood trough concentration above the recommended therapeutic range (>15 ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag Pty Ltd Clinical Trial, Study Director — Janssen-Cilag Pty Ltd

REFERENCES:
- [Derived] Campbell S, Hawley C, Irish A, Hutchison B, Walker R, Butcher BE, Ferrari P. Pre-transplant pharmacokinetic profiling and tacrolimus requirements post-transplant. Nephrology (Carlton). 2010 Oct;15(7):714-9. doi: 10.1111/j.1440-1797.2010.01351.x. PMID 21040167